CLINICAL TRIAL: NCT01413711
Title: An Open-Label, Single and Multiple Oral Dose Pharmacokinetic Study of Vigabatrin in Infants With Infantile Spasms
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13453A
Record Dates: First submitted 2011-06-17; First posted 2011-08-10 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Infantile Spasms
Keywords: IS; Pharmacokinetics; Area under the curve; Maximum plasma concentration; Time to maximum concentration
MeSH Terms: conditions — Spasms, Infantile | interventions — Vigabatrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vigabatrin (Experimental)
  Interventions: Drug: Vigabatrin

INTERVENTIONS:
Drug: Vigabatrin — Oral vigabatrin as a single 25 mg/kg dose on Days 1 and 5, 25 mg/kg twice a day (50 mg/kg daily dose, orally) on Days 2-4
  Other Names: Sabril®

SUMMARY:
The primary objective of the study is to evaluate vigabatrin pharmacokinetics (PK) in neonates receiving vigabatrin for infantile spasms (IS); and to determine the safety of vigabatrin.

ELIGIBILITY:
Inclusion Criteria:

* The patient's parent or legally authorized representative is able to read and understand the Patient Information Sheet and Informed Consent Form.
* The patient's legally authorized representative has signed the Informed Consent Form.
* The patient has IS, diagnosed according to the International League Against Epilepsy (ILAE) criteria.
* The patient is a full term (38 weeks gestation) male or female, aged >=1 month to <6 months at the time of enrollment.
* The patient's length and body weight for gestational age is >=5th and <=95th percentile, according to Centers for Disease Control and Prevention (CDC) Growth Charts.

Exclusion Criteria:

* The patient is currently being treated or has been previously treated with vigabatrin.
* The patient is a member of the site personnel's immediate family.
* The patient takes or has taken disallowed recent or concomitant medication or it is anticipated that the patient will require treatment with at least one of the disallowed concomitant medications during the study.
* The patient has a history of severe drug allergy or hypersensitivity, or known hypersensitivity to the investigational medicinal product (IMP) or the excipients (povodone/iodine) of the IMP.
* The patient has any other disorder for which the treatment takes priority over treatment of IS or is likely to interfere with study treatment or impair treatment compliance.
* The patient has been treated with any IMP within 30 days or 5 half lives (whichever is longer) prior to the Screening Visit.
* The patient has a disease or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.
* The patient has been diagnosed or is judged by the investigator to have anemia.
* The patient has been diagnosed or is judged by the investigator to have renal insufficiency.
* The patient's parent or legally authorized representative is, in the investigator's opinion, unlikely or unwilling to comply with the protocol or the patient is unsuitable for any reason.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Non-compartmental pharmacokinetic profile of vigabatrin after oral administrations in infants(>=1 and <6 months of age) | 24 hrs post dose on Day 1 and 12 hrs post dose on Day 5
  Serial blood for plasma generation will be collected on Days 1 and 5 and vigabatrin concenrations determined to the determine the pharmacokinetic profile of vigabatrin

SECONDARY OUTCOMES:
To determine the safety of vigabatrin following oral dose administrations in infants (>=1 and <6 months of age) | Safety collected throughout the 5-day study
  Safety and tolerability parameters such as adverse events, clinical safety laboratory tests and vital signs will be summarised using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com